CLINICAL TRIAL: NCT05619172
Title: A Phase 2, Open-label, Single-arm, Multicenter Study to Evaluate the Efficacy and Safety of SOT101 in Combination With Cetuximab in Patients With RAS Wild-type Colorectal Cancer
Brief Title: A Study of Nanrilkefusp Alfa (SOT101) in Combination With Cetuximab to Evaluate the Efficacy and Safety in Patients With Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lack of efficacy shown at the time of the interim analysis.
Sponsor: SOTIO Biotech AG (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SC105; AURELIO-05 (Other: SOTIO Biotech AG); 2022-001527-32 (EudraCT Number)
Record Dates: First submitted 2022-11-01; First posted 2022-11-16 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
Keywords: SOT101; SO-C101; Cetuximab; Colorectal cancer; AURELIO-05; Nanrilkefusp alfa
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Intervention Model Description: Study SC105 (AURELIO-05) was a phase 2, open-label, single-arm, multicenter study of nanrilkefusp alfa in combination with cetuximab with an initial safety run-in with 3+3 safety cohorts. Two safety cohorts were implemented. The main cohort was not opened.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nanrilkefusp alfa 9 µg/kg and cetuximab (Experimental): Participants were treated with 9 µg/kg of nanrilkefusp alfa in combination with cetuximab. Nanrilkefusp alfa treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 2 (±1 day), day 8 (±1 day), and day 9 (±1 day) of each 21-day cycle. Cetuximab treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 8 (±1 day), and day 15 (±1 day) of each 21-day cycle; on day 1 and day 8, cetuximab infusion started within 30 minutes after nanrilkefusp alfa administration.
  Interventions: Drug: Nanrilkefusp alfa; Drug: Cetuximab
- Nanrilkefusp alfa 12 µg/kg and cetuximab (Experimental): Participants were treated with 12 µg/kg of nanrilkefusp alfa in combination with cetuximab. Nanrilkefusp alfa treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 2 (±1 day), day 8 (±1 day), and day 9 (±1 day) of each 21-day cycle. Cetuximab treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 8 (±1 day), and day 15 (±1 day) of each 21-day cycle; on day 1 and day 8, cetuximab infusion started within 30 minutes after nanrilkefusp alfa administration.
  Interventions: Drug: Nanrilkefusp alfa; Drug: Cetuximab

INTERVENTIONS:
Drug: Nanrilkefusp alfa — Subcutaneous (SC) injection
Drug: Cetuximab — Intravenous (IV) infusion via peripheral or central venous line

SUMMARY:
The primary objective of the study is to estimate the antitumor efficacy of nanrilkefusp alfa (SOT101) in combination with cetuximab in RAS wild-type colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

*Type of patients*

1. ≥18 years of age on the day of signing informed consent
2. Ability to understand and sign written informed consent to participate in the study
3. Provides written informed consent for the study
4. Life expectancy >6 months

   *Disease characteristics*
5. Histologically or cytologically confirmed advanced and/or metastatic colorectal cancer
6. RAS wild type as confirmed by:

   * locally performed US Food and Drug Administration (FDA)-approved test or an experienced local laboratory using validated test methods for the detection, based on tumor biopsy or
   * locally performed ctDNA assessment including at least mutations in exon 2 (G12D, G12V, G12C, G12S, G12A, G12R, G13D) and determined by a laboratory using validated test methods
   * samples must be taken within 3 months prior to first study administration
7. Patients who are relapsed/refractory or intolerant to prior treatment with irinotecan- and oxaliplatin-containing chemotherapy
8. Have at least one measurable lesion according to RECIST 1.1
9. Eastern Cooperative Oncology Group (ECOG) performance score 0-2
10. Must have recovered from all AEs due to previous therapies to grade ≤1 toxicity (excluding alopecia)

    *Organ function: Have adequate organ function as defined below. Specimens must be collected within 7 days prior to the start of study treatment.*
11. Hematology:

    11.1. Absolute neutrophil count ≥1,500/µL 11.2. Platelets ≥100,000/µL 11.3. Hemoglobin ≥9.0 g/dL (criteria must be met without packed red blood cell transfusion within the prior 2 weeks; patients can be on stable dose of erythropoietin [≥3 months])
12. Renal function: Creatinine clearance rate ≥50 mL/min as calculated using Cockcroft-Gault equation
13. Hepatic function: ALT/AST ≤2.5× upper limit of normal (ULN) and total bilirubin ≤2×ULN in patients without liver metastasis (benign hereditary hyperbilirubinemias, e.g., Gilbert's syndrome, are permitted if total bilirubin <3 mg/dL). In patients with liver metastasis, ALT/AST ≤5×ULN is allowed but total bilirubin must be ≤2×ULN.
14. Prothrombin time and activated partial thromboplastin time ≤1.5×ULN

    *Hepatitis*
15. A locally performed hepatitis B (HBV) test is required during screening. Patients who are HBV surface antigen positive are eligible if they have received HBV anti-viral therapy for at least 4 weeks and have undetectable HBV viral load before study entry (ICF signature). Patients should remain on anti-viral therapy throughout study treatment and follow local guidelines for HBV anti-viral therapy post completion of study treatments.
16. A locally performed hepatitis C (HCV) test is required during screening. Patients with history of HCV infection are eligible if HCV viral load is undetectable at screening. Patients must have completed anti-viral therapy at least 4 weeks before study entry (ICF signature).

    *Special requirements for contraception*
17. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and one of the following conditions applies:

    17.1. Not a woman of childbearing potential (WOCBP). A WOCBP is defined as fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single follicle stimulating hormone measurement is insufficient.

    17.2. A WOCBP who agrees to use a highly effective contraceptive method during the treatment period and for at least 60 days after the last dose of cetuximab or at least 30 days after last dose of nanrilkefusp alfa, whichever is later. A WOCBP can only be included after a negative serum pregnancy test at screening within 7 days before day 1 of cycle 1.
18. Male patients must agree to use a condom during the treatment period and for at least 60 days after the last dose of cetuximab or at least 30 days after last dose of nanrilkefusp alfa, whichever is later.

Exclusion Criteria:

*Prior/concomitant therapy*

1. Prior exposure to drugs that are agonists of IL-2 or IL-15
2. Therapy with cetuximab within 3 months prior to ICF signature or patients who had progressive disease as best response to prior cetuximab-containing regimen
3. Prior systemic anti-cancer therapies, including investigational agents before study entry (ICF signature):

   3.1. Less than 3 weeks or 5 half lives (whichever shorter) for anti-cancer treatments 3.2. Less than 4 weeks from major surgeries and not recovered adequately from the procedure and/or any complications from the surgery
4. Has received more than 4 prior lines of systemic anticancer treatment
5. Has received prior radiotherapy within 2 weeks of the start of study treatments. A 1-week radiation-free period is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system disease. Patients must have recovered from all radiation-related toxicities and not require corticosteroids.
6. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study treatments

   *Prior/concurrent clinical study experience*
7. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 3 weeks or 5 half lives (whichever longer) before study entry (ICF signature). Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 3 weeks or 5 half lives (whichever longer) after the last dose of the previous investigational agent.

   *Medical conditions*
8. Patients with known BRAF mutations
9. Clinically significant cardiac abnormalities including prior history of any of the following:

   9.1. Cardiomyopathy, with left ventricular ejection fraction lower than the lower limit of the institutional normal range at screening 9.2. Congestive heart failure of New York Heart Association grade ≥2 9.3. History of clinically significant (i.e., active) atherosclerotic cardiovascular disease, specifically myocardial infarction, unstable angina, cerebrovascular accident within 6 months prior to the first dose of study treatments, and any history of coronary heart disease and clinically significant peripheral and/or carotid artery disease 9.4. Prolongation of QTcF >450 msec; history or family history of congenital long QT syndrome 9.5. Uncontrolled cardiac arrhythmia requiring medication
10. Uncontrolled hypertension defined as systolic blood pressure >160 mmHg, diastolic blood pressure >110 mmHg. Patients with uncontrolled hypertension should be medically managed on a stable regimen to control hypertension prior to study entry (ICF signature).
11. Has a clinical diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatments. Systemic steroid pretreatment prior to cetuximab infusion according to local guidelines is permitted.
12. History of or serology positive for HIV. A locally performed HIV test is required during screening.
13. Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Patients with basal cell carcinoma of the skin or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are eligible.
14. Has known active central nervous system metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks confirmed during screening.
15. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
16. Has an active infection requiring systemic therapy
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
18. Has a known psychiatric or substance abuse disorder that would interfere with the patient's ability to cooperate with the requirements of the study
19. History of hypersensitivity to any component of cetuximab or to compounds of similar biological or chemical composition of nanrilkefusp alfa and/or the excipients contained in the study drug formulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-06-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (2):
  - Grand Hopital de Charleroi - Hopital Notre Dame, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
- France (2):
  - Institut Bergonié, Bordeaux
  - Hopital Foch, Suresnes
- Spain (4):
  - Vall d'Hebron Institut d'Oncologia (VHIO), Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - HM Universitario Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Safety Cohort 1
Arm/Group | Nanrilkefusp Alfa 9 µg/kg and Cetuximab | Nanrilkefusp Alfa 12 µg/kg and Cetuximab
Started | 14 | 0
Completed | 0 | 0
Not Completed | 14 | 0
Not completed — Death | 7 | 0
Not completed — Study terminated by sponsor | 7 | 0
Period: Safety Cohort 2
Arm/Group | Nanrilkefusp Alfa 9 µg/kg and Cetuximab | Nanrilkefusp Alfa 12 µg/kg and Cetuximab
Started | 0 | 2
Completed | 0 | 0
Not Completed | 0 | 2
Not completed — Death | 0 | 1
Not completed — Study terminated by sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Nanrilkefusp Alfa and Cetuximab: Participants were treated with nanrilkefusp alfa (safety cohort 1: 14 participants with 9 µg/kg nanrilkefusp alfa; safety cohort 2: 2 participants with 12 µg/kg nanrilkefusp alfa) in combination with cetuximab. Per statistical considerations outlined in the trial Protocol and Statistical Analysis Plan, all patients were analyzed within pre-specified populations across the entire trial. There was no plan to analyze cohorts separately; therefore, results are presented in aggregate. The trial was a single-arm design, not a classic dose-escalation study, as the RP2D (12 µg/kg) had been established in a prior trial (NCT04234113). The 9 µg/kg dose was a safety cohort allowing one-way crossover to 12 µg/kg.
  Nanrilkefusp alfa treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 2 (±1 day), day 8 (±1 day), and day 9 (±1 day) of each 21-day cycle. Cetuximab treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 8 (±1 day), and day 15 (±1 day) of each 21-day cycle; on day 1 and day 8, cetuximab infusion started within 30 minutes after nanrilkefusp alfa administration.
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  Belgium | 7
  France | 3
  Spain | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1)
Description: Objective response rate according to RECIST 1.1 was defined as the proportion of participants with complete response according to RECIST 1.1 or partial response according to RECIST 1.1 for target lesions and assessed by CT/MRI. Participants with missing data were considered non-responders.
Time Frame: Day 1 up to approximately 1 year 2 months
Population: Per statistical considerations outlined in the trial Protocol and Statistical Analysis Plan, all patients were analyzed within pre-specified populations across the entire trial. There was no plan to analyze cohorts separately; therefore, results are presented in aggregate. The trial was a single-arm design, not a classic dose-escalation study, as the RP2D (12 µg/kg) had been established in a prior trial (NCT04234113). The 9 µg/kg dose was a safety cohort allowing one-way crossover to 12 µg/kg.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Nanrilkefusp Alfa and Cetuximab: Participants were treated with nanrilkefusp alfa in combination with cetuximab. Safety cohort 1: 14 participants were treated with 9 µg/kg nanrilkefusp alfa; safety cohort 2: 2 participants were treated with 12 µg/kg nanrilkefusp alfa. Nanrilkefusp alfa treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 2 (±1 day), day 8 (±1 day), and day 9 (±1 day) of each 21-day cycle. Cetuximab treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 8 (±1 day), and day 15 (±1 day) of each 21-day cycle; on day 1 and day 8, cetuximab infusion started within 30 minutes after nanrilkefusp alfa administration.
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
percentage of participants | 0 [0 to 20.591]

2. Secondary Outcome: Objective Response Rate According to RECIST for Immune-based Therapeutics (iRECIST)
Description: Objective response rate according to iRECIST was defined as the proportion of participants with complete response according to iRECIST or partial response according to iRECIST for target lesions and assessed by CT/MRI. Participants with missing data were considered non-responders.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
percentage of participants | 0 [0 to 20.591]

3. Secondary Outcome: Best Overall Response According to RECIST 1.1: Number of Participants With Complete Response
Description: The best overall response according to RECIST 1.1 was defined as the best response from the start of study treatment until the first documented disease progression, death, or start of new anti-cancer therapy for target lesions and assessed by CT/MRI.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 0

4. Secondary Outcome: Best Overall Response According to RECIST 1.1: Number of Participants With Partial Response
Description: as for outcome 3
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 0

5. Secondary Outcome: Best Overall Response According to RECIST 1.1: Number of Participants With Stable Disease
Description: The best overall response according to RECIST 1.1 was defined as the best response from the start of study treatment until the first documented disease progression, death, or start of new anti-cancer therapy for target lesions and assessed by CT/MRI. Stable disease according to RECIST 1.1 had to last at least 6 weeks from the start of study treatment. If not, at least 1 follow-up scan was required to declare stable disease.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 6

6. Secondary Outcome: Best Overall Response According to RECIST 1.1: Number of Participants With Progressive Disease
Description: as for outcome 3
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 7

7. Secondary Outcome: Best Overall Response According to iRECIST: Number of Participants With Complete Response
Description: The best overall response according to iRECIST was defined as the best response from the start of study treatment until the first documented disease progression, death, or start of new anti-cancer therapy for target lesions and assessed by CT/MRI.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 0

8. Secondary Outcome: Best Overall Response According to iRECIST: Number of Participants With Partial Response
Description: as for outcome 7
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 0

9. Secondary Outcome: Best Overall Response According to iRECIST: Number of Participants With Stable Disease
Description: The best overall response according to iRECIST was defined as the best response from the start of study treatment until the first documented disease progression, death, or start of new anti-cancer therapy for target lesions and assessed by CT/MRI. Stable disease according to iRECIST had to last at least 6 weeks from the start of study treatment. If not, at least 1 follow-up scan was required to declare stable disease.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 6

10. Secondary Outcome: Best Overall Response According to iRECIST: Number of Participants With Unconfirmed Progressive Disease
Description: as for outcome 7
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 5

11. Secondary Outcome: Best Overall Response According to iRECIST: Number of Participants With Confirmed Progressive Disease
Description: as for outcome 7
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 2

12. Secondary Outcome: Duration of Response According to RECIST 1.1
Description: Duration of response according to RECIST 1.1 was defined as time to disease progression for participants with partial response or complete response according to RECIST 1.1.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: As outlined in the trial Protocol and Statistical Analysis Plan, patients were analyzed within pre-specified populations across the trial. There was no plan to analyze cohorts separately; results are presented in aggregate. The trial was a single-arm design, not a dose-escalation study; the RP2D (12 µg/kg) was established in a prior trial (NCT04234113). The 9 µg/kg dose was a safety cohort with one-way crossover to 12 µg/kg.
  No participant had a PR or CR per RECIST; DoR data were not collected.
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 0

13. Secondary Outcome: Duration of Response According to iRECIST
Description: Duration of response according to iRECIST was defined as time to disease progression for participants with partial response or complete response according to iRECIST.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: As outlined in the trial Protocol and Statistical Analysis Plan, patients were analyzed within pre-specified populations across the trial. There was no plan to analyze cohorts separately; results are presented in aggregate. The trial was a single-arm design, not a dose-escalation study; the RP2D (12 µg/kg) was established in a prior trial (NCT04234113). The 9 µg/kg dose was a safety cohort with one-way crossover to 12 µg/kg.
  No participant had a PR or CR per iRECIST; DoR data were not collected
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 0

14. Secondary Outcome: Clinical Benefit Rate According to RECIST 1.1
Description: Clinical benefit rate according to RECIST 1.1 was defined as the number of partial responses, complete responses, and stable disease according to RECIST 1.1. Stable disease had to last at least 6 weeks from the start of study treatment. If not, at least 1 follow-up scan was required to declare stable disease. Participants with missing data were considered non-responders.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
percentage of participants | 37.5 [15.198 to 64.565]

15. Secondary Outcome: Clinical Benefit Rate According to iRECIST
Description: Clinical benefit rate according to iRECIST was defined as the number of partial responses, complete responses, and stable disease according to iRECIST. Stable disease had to last at least 6 weeks from the start of study treatment. If not, at least 1 follow-up scan was required to declare stable disease. Participants with missing data were considered non-responders.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
percentage of participants | 37.5 [15.198 to 64.565]

16. Secondary Outcome: Progression-free Survival According to RECIST 1.1
Description: Progression-free survival according to RECIST 1.1 was defined as the time from the first day of study treatment to the first date of radiological disease progression according to RECIST 1.1 or death.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
months | 2.7 [1.05 to 3.94]

17. Secondary Outcome: Progression-free Survival According to iRECIST
Description: Progression-free survival according to iRECIST was defined as the time from the first day of study treatment to the first date of radiological disease progression according to iRECIST or death.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
months | 2.7 [1.05 to 3.94]

18. Secondary Outcome: Time to Response According to RECIST 1.1
Description: Time to response according to RECIST 1.1 was defined as the time from the first day of study treatment to the first date of partial response or complete response according to RECIST 1.1. Participants with missing data were censored at the last assessment date, date of death, or date of eligibility (for incomplete or missing baseline tumor assessments), whichever occurred last.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
months | 0 [0 to 0]

19. Secondary Outcome: Time to Response According to iRECIST
Description: Time to response according to iRECIST was defined as the time from the first day of study treatment to the first date of partial response or complete response according to iRECIST. Participants with missing data were censored at the last assessment date, date of death, or date of eligibility (for incomplete or missing baseline tumor assessments), whichever occurred last.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
months | 0 [0 to 0]

20. Secondary Outcome: Time to Progression According to RECIST 1.1
Description: Time to progression according to RECIST 1.1 was defined as the time from the first day of study treatment to the first date of radiological disease progression according to RECIST 1.1.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
months | 2.8 [1.35 to 3.94]

21. Secondary Outcome: Time to Progression According to iRECIST
Description: Time to progression according to iRECIST was defined as the time from the first day of study treatment to the first date of radiological disease progression according to iRECIST.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
months | 2.8 [1.35 to 3.94]

22. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: A treatment-emergent adverse event is defined as an adverse event that started or worsened at or after the start of study treatment.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 16

23. Secondary Outcome: Number of Participants With Clinical Laboratory Test Abnormalities (Coagulation, Hematology, Clinical Chemistry and Urinalysis)
Description: The following laboratory parameters will be assessed:
  Coagulation: prothrombin time, activated partial thromboplastin time, international normalized ratio, D-dimer, and fibrinogen
  Hematology: hemoglobin, glycated hemoglobin at screening, hematocrit, red blood cell count, reticulocytes, white blood cell count (with full differentiation), absolute lymphocyte count, and platelet count
  Clinical chemistry: Na, K, Cl, phosphate, Mg, Ca, albumin, total protein, ALT, AST, bilirubin (direct, total), alkaline phosphatase, lactate dehydrogenase, creatinine clearance calculated by the Cockcroft-Gault formula, creatinine, glucose (preferably fasting), urea or blood urea nitrogen, cholesterol, triglyceride, C-reactive protein, uric acid, amylase, and lipase
  Urinalysis: pH, glucose, protein, bilirubin, urobilinogen. Microscopic examination (mandated only if clinically indicated): red blood cell count, white blood cell count, epithelial cells, bacteria
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 11

24. Secondary Outcome: Number of Participants With Vital Signs Abnormalities
Description: The following vital signs parameters will be assessed:
  Blood pressure (systolic and diastolic, after ≥5 minutes of rest), body temperature, and heart rate
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 11

25. Secondary Outcome: Number of Participants With Electrocardiography Abnormalities
Description: Standard 12-lead electrocardiography was evaluated locally.
Time Frame: Day 1 up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 1

26. Secondary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: The following adverse events as per NCI CTCAE version 5.0 were considered dose-limiting toxicities:
  * All grade 5 events not clearly related to disease progression or any other causes
  * Any grade 3 or higher non-hematologic toxicity regardless of duration; exceptions:
    * Grade 3 nausea, vomiting, or diarrhea that could be controlled within 72 hours
    * Grade 3 fatigue lasting less than 5 days
    * Grade 3 or higher correctable electrolyte abnormalities lasting less than 72 hours and not associated with clinical complications
    * Grade 3 or higher serum amylase or lipase not associated with clinical manifestations of pancreatitis
    * Grade 3 AST or ALT increase or grade 3 blood bilirubin increase lasting 5 days or less
  * Hy's law cases
  * Hematologic DLTs:
    * Grade 4 decreased neutrophil count or decreased platelet count lasting more than 7 days
    * Febrile neutropenia
    * Grade 3 or higher decreased platelet count with bleeding
Time Frame: Through Cycle 1 (21 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 6
Participants | 0

27. Secondary Outcome: Characterization of Area Under the Curve of Nanrilkefusp Alfa
Description: At 9 µg/kg nanrilkefusp alfa on Day 1 of Cycle 1
Time Frame: Day 1 of Cycle 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h*ng/mL
Groups:
- Nanrilkefusp Alfa and Cetuximab: Participants were treated with 9 µg/kg nanrilkefusp alfa in combination with cetuximab. Nanrilkefusp alfa treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 2 (±1 day), day 8 (±1 day), and day 9 (±1 day) of each 21-day cycle. Cetuximab treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 8 (±1 day), and day 15 (±1 day) of each 21-day cycle; on day 1 and day 8, cetuximab infusion started within 30 minutes after nanrilkefusp alfa administration.
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 13
h*ng/mL | 37.1 [21.8 to 88.5]

28. Secondary Outcome: Characterization of Maximum Concentration of Nanrilkefusp Alfa on Day 1 of Cycle 1
Description: At 9 µg/kg nanrilkefusp alfa
Time Frame: Day 1 of Cycle 1
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 13
ng/mL | 3.56 [1.45 to 6.78]

29. Secondary Outcome: Characterization of Time to Maximum Concentration of Nanrilkefusp Alfa on Day 1 of Cycle 1
Description: At 9 µg/kg nanrilkefusp alfa
Time Frame: Day 1 of Cycle 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 13
hours | 6.21 [2.03 to 22.8]

30. Secondary Outcome: Characterization of Pre-dose Concentration of Nanrilkefusp Alfa on Day 1 of Cycle 1
Description: At 9 µg/kg nanrilkefusp alfa
Time Frame: Day 1 of Cycle 1
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 13
ng/mL | 0.404 [0.178 to 1.50]

31. Secondary Outcome: Incidence of Treatment-induced Anti-drug Antibodies Against Nanrilkefusp Alfa
Description: At 9 µg/kg and 12 µg/kg nanrilkefusp alfa
Time Frame: Day 1 until 30 (±2) days after the last dose of nanrilkefusp alfa, up to approximately 1 year 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nanrilkefusp Alfa and Cetuximab
Number analyzed (Participants) | 16
Participants | 5

ADVERSE EVENTS:
Time Frame: Adverse events: from the start of study treatment to 90 days after the end of study treatment up to approximately 1 year 5 months; related serious adverse events: collected beyond 90 days after the end of study treatment up to approximately 1 year 5 months; deaths: consent signature to study end up to approximately 1 year 5 months
Description: Only treatment-emergent adverse events were analyzed (see the definition above); the tables include information on treatment-emergent adverse events, serious treatment-emergent adverse events, and all deaths; causality was assessed by investigators. The two safety cohorts are not described separately due to the small number of participants in safety cohort 2.
Groups:
- Nanrilkefusp Alfa and Cetuximab 9 µg/kg (Safety Cohort 1): Participants were treated with nanrilkefusp alfa in combination with cetuximab. 14 participants were treated with 9 µg/kg nanrilkefusp alfa. Nanrilkefusp alfa treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 2 (±1 day), day 8 (±1 day), and day 9 (±1 day) of each 21-day cycle. Cetuximab treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 8 (±1 day), and day 15 (±1 day) of each 21-day cycle; on day 1 and day 8, cetuximab infusion started within 30 minutes after nanrilkefusp alfa administration.
- Nanrilkefusp Alfa and Cetuximab 12 µg/kg (Safety Cohort 2): Participants were treated with nanrilkefusp alfa in combination with cetuximab. 2 participants were treated with 12 µg/kg nanrilkefusp alfa. Nanrilkefusp alfa treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 2 (±1 day), day 8 (±1 day), and day 9 (±1 day) of each 21-day cycle. Cetuximab treatment was administered on day 1 (from cycle 2 onwards, ±1 day), day 8 (±1 day), and day 15 (±1 day) of each 21-day cycle; on day 1 and day 8, cetuximab infusion started within 30 minutes after nanrilkefusp alfa administration.
Arm/Group | Nanrilkefusp Alfa and Cetuximab 9 µg/kg (Safety Cohort 1) | Nanrilkefusp Alfa and Cetuximab 12 µg/kg (Safety Cohort 2)
All-Cause Mortality (participants affected / at risk) | 7/14 | 1/2
Serious Adverse Events (participants affected / at risk) | 7/14 | 1/2
Other Adverse Events (participants affected / at risk) | 14/14 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nanrilkefusp Alfa and Cetuximab 9 µg/kg (Safety Cohort 1) (N=14) | Nanrilkefusp Alfa and Cetuximab 12 µg/kg (Safety Cohort 2) (N=2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Disease progression (General disorders) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nanrilkefusp Alfa and Cetuximab 9 µg/kg (Safety Cohort 1) (N=14) | Nanrilkefusp Alfa and Cetuximab 12 µg/kg (Safety Cohort 2) (N=2)
Hypotension (Vascular disorders) | 2 (4) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 10 (12) | 1 (1)
Pyrexia (General disorders) | 8 (26) | 2 (2)
Injection site reaction (General disorders) | 7 (7) | 0 (0)
Chills (General disorders) | 2 (6) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 5 (8) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 8 (11) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 1 (2) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (7) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results will be published and/or presented at scientific meetings in their totality in a timely manner. Any formal publication of clinical trial results will be a collaborative effort between the sponsor and the investigator(s). All manuscripts or abstracts will be reviewed and approved in written by the sponsor before submission. The sponsor may request a delay in publication if there are important intellectual property concerns.

DOCUMENTS (2):
  • Study Protocol (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT05619172/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT05619172/SAP_001.pdf